CLINICAL TRIAL: NCT01320930
Title: Early Detection and Rehabilitation of Subjects With COPD - Rehabilitation in Moderate COPD
Brief Title: Rehabilitation in Subjects With Moderate Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government); Danish Lung Association (Other); Sygekassernes Helsefond (Other)
Responsible Party: Vibeke Backer, professor, MD., The Department of Respiratory Medicine, L, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TORKOL1
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Effect of Pulmonary rehabilitation.; Exercise capacity; Quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary rehabilitation (Active Comparator): A standardized 7 week rehabilitation program, including physical training and education.
  Interventions: Behavioral: Pulmonary rehabilitation
- Control (Placebo Comparator): Conventional care
  Interventions: Behavioral: conventional care

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation
  Arms: Pulmonary rehabilitation
Behavioral: conventional care
  Arms: Control

SUMMARY:
The study is a single-center randomized, unblinded, placebo-controlled study to investigate the effect of pulmonary rehabilitation in subjects with moderate chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of moderate COPD.
2. Motivation for Pulmonary rehabilitation.

Exclusion Criteria:

1. Comorbidity contraindicating rehabilitation.
2. Participation in pulmonary rehabilitation within the last year.
3. Cognitive disorders limiting the ability to participate in physical training and education sessions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-01; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)